CLINICAL TRIAL: NCT01965171
Title: Transfusional Iron Overload Among Leukemia Survivors
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: TRIALS
Record Dates: First submitted 2013-10-11; First posted 2013-10-18 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Acute Lymphocytic Leukemia; Acute Myeloid Leukemia
Keywords: hematologic malignancy; iron overload; magnetic resonance imaging; childhood cancer survivors
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Hematologic Neoplasms; Iron Overload

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Red cell transfusions are an important part of supportive cancer therapy. The iron in the transfused blood may build up in the body since the human body has no way to get rid of extra iron. Iron tends to build up in the liver and the heart muscle. It is unknown if iron build-up is present many years after completing cancer therapy. It is also not known if extra iron causes harm to internal organs. Researchers at St. Jude Children's Research Hospital (SJCRH) want to understand if iron build-up (called "iron overload") exists in survivors of leukemia. They also want to know if iron overload can cause injury to your organs if it is present.

Liver iron accumulation has been documented in childhood cancer survivors, however, it is not known if iron associated organ toxicity is contributing to the long-term morbidity that has been well documented among these survivors. This study will investigate the prevalence of iron overload and the association of tissue iron burden with markers of organ dysfunction in leukemia survivors. This study will determine the prevalence of iron overload among long-term leukemia survivors that underwent blood transfusion. This study will use blood and magnetic resonance imaging (MRI) testing to determine iron overload of specified organs. Understanding the prevalence of iron overload could impact surveillance practices in leukemia survivors.

PRIMARY OBJECTIVE:

* To determine the prevalence of iron overload in the liver [liver iron concentration (LIC) >3mg/g using R2* MRI measurements] and in the heart (T2* <20 ms) among long-term leukemia survivors transfused with ≥50ml/kg of packed red blood cells.

SECONDARY OBJECTIVES:

* To examine the relationship between hepatic, cardiac, and endocrine dysfunction and transfusionally acquired iron overload as defined by R2* and T2* MRI among survivors of pediatric leukemias.
* To investigate the association between serum ferritin, transferrin saturation, non-transferrin-bound iron, and hepcidin measurements with R2* and T2* MRI-defined iron overload.

DETAILED DESCRIPTION:
Participants will have blood work drawn after an overnight fast during a routine clinic visit. They will also have an electrocardiogram (EKG) and echocardiogram (ECHO) which are often a required part of their annual visit. Magnetic resonance imaging (MRI) exams of the heart, liver, and surrounding abdominal organs will be done on all participants using a method of scanning that involves a closer study of these organs (called R2* MRI).

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of ALL or AML that was treated at SJCRH with conventional chemotherapy.
* At time of enrollment survivors should be > 5 and < 10 years from diagnosis of primary cancer.
* A packed red blood cell transfusion history of ≥50 ml/kg.

Exclusion Criteria:

* Undergoing active cancer therapy for relapse or subsequent malignant neoplasm
* History of hematopoietic stem cell transplant (HSCT)
* A known disorder of iron regulation such as hereditary hemochromatosis
* Any contraindication to undergoing an MRI, such as the presence of ferromagnetic material in the body
* If patient is an adult (18 years or over), does require IV sedation or anxiolytic to undergo MRI
* Positive pregnancy test, or known ongoing pregnancy

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will have been treated at SJCRH for acute lymphoblastic leukemia (ALL) or acute myeloid leukemia (AML) and would have received ≥50 ml/kg of packed red blood cells during their treatment.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2013-10-18 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Proportion of iron overload | On day of enrollment
  Iron overload will be measured by R2*MRI in the liver and T2* in the heart and is defined as R2*MRI value > 3 mg/g and/or T2* MRI <20ms.

SECONDARY OUTCOMES:
Relationship between hepatic, cardiac, and endocrine dysfunction and transfusionally-acquired iron overload | On day of enrollment
  Fisher's Exact test will be performed to examine the relationship of organ dysfunction and iron overload. Then the logistic regression model will be built to evaluate the effect of the iron overload defined by R2* and T2* MRI on the risk of organ dysfunction, respectively, while controlling for the effects of craniospinal radiation and chemotherapeutic agents.
Association between serum ferritin, transferrin saturation, non-transferrin-bound iron, and hepcidin measurements with R2* and T2* MRI-defined iron overload | On day of enrollment
  Logistic regression model will be used to evaluate the association of iron overload status and the above four iron test measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Hankins, MD, MS, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols